CLINICAL TRIAL: NCT00345202
Title: Short Term Effects of HMG-CoA Reductase Inhibition (Atorvastatin)on Renal Hemodynamics, Tubular Function and Vasoactive Hormones on Healthy Subjects.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MED.RES.HOS.2004.02.LP
Record Dates: First submitted 2006-06-24; First posted 2006-06-27 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Healthy
Keywords: HMG-COA reductase inhibition; GFR; RPF; FE; CL
MeSH Terms: interventions — Atorvastatin

INTERVENTIONS:
Drug: HMG-CoA reductase inhibition (atorvastatin)

SUMMARY:
We wanted to test the shortterm effects of HMG-CoA reductase inhibition (atorvastatin) on renal hemodynamics, renal tubular function and vasoactive hormones on healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Both men and women
* Age: Between 20-50
* BMI<30

Exclusion Criteria:

* Cl. signs or history of disease of heart, lungs, kidneys or endocrine organs.
* Abnormal lab. tests( haemoglobin, pl. sodium, pl. potassium, pl.creatinine, pl.bilirubin, pl.ALAT, pl. cholesterol, blood glucose)
* Albuminuria or glucosuria
* Cancer
* Art. hypertension
* Alcohol abuse
* Med. treatment, except oral contraceptives
* Pregnancy or breast feeding
* Blood donation less than 1 month before study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2004-09; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
GFR
RPF
FEna
FELi
CLna
CLli

CONTACTS AND LOCATIONS:
Overall Officials: Erling B. Pedersen, Professor, Study Chair — Holstebro Sygehus
Locations (1):
- Medical research unit, Department of medicin, Holstebro Sygehus, Holstebro, Ringkøbing Countie, Denmark